CLINICAL TRIAL: NCT01990482
Title: Influence of Coffee Intake on Postoperative Bowel Function After Comprehensive Staging Surgery for Gynecological Malignancies: A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Medical Doctor, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gungorduk15
Record Dates: First submitted 2013-11-10; First posted 2013-11-21 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2013-11

CONDITIONS: Ilues
MeSH Terms: interventions — Water

ARMS (2):
- coffee (Experimental): coffee
  Interventions: Dietary Supplement: caffe; Dietary Supplement: Water
- water group (Placebo Comparator): water
  Interventions: Dietary Supplement: caffe; Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: caffe
Dietary Supplement: Water

SUMMARY:
A delay in the return of normal bowel function with the passage of flatus and feces is one of the most important factors affecting early recovery and discharge in patients undergoing open complete staging surgery for gynecological malignancies. A prolonged hospital stay increases the risk of hospital-acquired infections, deep vein thrombosis, pulmonary compromise and total hospital costs.

The aim of this study was to assess the effectiveness of coffee intake on postoperative bowel function in patients undergoing abdominal complete staging surgery for gynecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Female patients preparing for complete surgical staging for malignant gynecologic disease such as endometrial cancer, cervix cancer and ovarian cancerwere assessed for eligibility. Exclusion Criteria: Exclusion criteria for the study
* included thyroid diseases,
* inflammatory bowel disease,
* complaints of chronic constipation (defined as two or fewer bowel movements per week),
* a history of prior abdominal bowel surgery, abdominal radiation, neoadjuvant chemotherapy,
* need for intensive care more that 24 hpostoperatively,
* nasogastric tube drainage beyond the first postoperative morning,
* bowel anastomosis and upper abdominalmultivisceral surgical approaches in relation to the debulking surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
time to first flatus | within the first 30 days after surgery
  hours from end of operation to first flatus pass time

SECONDARY OUTCOMES:
time to tolerance diet | within the first 30 days after surgery
  time to end of the surgery until the first solid diet intake without vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Education Research Hospital, Izmir, Tepecik, Turkey (Türkiye)